CLINICAL TRIAL: NCT03885830
Title: Preliminary Evaluation of TKI Exposure-response Relationships in Real World Patients (RWPs) With Chronic Myelogenous Leukemia (CML)
Brief Title: Precision Dosing of Tyrosine Kinase Inhibitors in CML Patients
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1906; 18-2424 (Other: University of North Carolina IRB)
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: CML, Chronic Phase; CML (Chronic Myelogenous Leukemia; CML - Philadelphia Chromosome; Chronic Myeloid Leukemia; Chronic Myeloid Leukemia, Chronic Phase
Keywords: Observational; Bosutinib; Dasatinib; Nilotinib; Imatinib; Chronic Myeloid Leukemia; CML; Pharmacokinetics
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib; Dasatinib; Imatinib Mesylate; nilotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For all study subjects, two blood samples will be taken at each study visit. These samples will be used to quantify TKI concentrations in the plasma. Later, the TKI concentration/time information will be used in PK analyses that will estimate clearance and exposure. Additionally, during the subject's first study, an additional blood sample will be obtained to isolate DNA for NGS. Throughout the study, all blood samples will be collected by a phlebotomist or nurse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Bosutinib: Subjects who have been prescribed or administered bosutinib (Bosulif) for treatment of chronic-phase CML for less than 12 months.
  Interventions: Drug: Bosutinib
- Dasatinib: Subjects who have been prescribed or administered dasatinib (Sprycel) for treatment of chronic-phase CML for less than 12 months.
  Interventions: Drug: Dasatinib
- Imatinib: Subjects who have been prescribed or administered imatinib (Gleevec) for treatment of chronic-phase CML for less than 12 months.
  Interventions: Drug: Imatinib
- Nilotinib: Subjects who have been prescribed or administered nilotinib (Tasigna) for treatment of chronic-phase CML for less than 12 months.
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Bosutinib — Subjects will be enrolled into this group if they are receiving bosutinib per standard of care. This is an observational study and no interventions will be made.
  Other Names: Bosulif
  Groups: Bosutinib
Drug: Dasatinib — Subjects will be enrolled into this group if they are receiving dasatinib per standard of care. This is an observational study and no interventions will be made.
  Other Names: Sprycel
  Groups: Dasatinib
Drug: Imatinib — Subjects will be enrolled into this group if they are receiving imatinib per standard of care. This is an observational study and no interventions will be made.
  Other Names: Gleevec
  Groups: Imatinib
Drug: Nilotinib — Subjects will be enrolled into this group if they are receiving nilotinib per standard of care. This is an observational study and no interventions will be made.
  Other Names: Tasigna
  Groups: Nilotinib

SUMMARY:
The purpose of this prospective, single-institution observational study is to evaluate associations between the pharmacokinetic (PK) parameters for tyrosine kinase inhibitors (TKIs) used to treat chronic phase chronic myeloid leukemia (CML) and clinical outcomes for up to 12 months. The study aims to identify associations between TKI clearance and/or exposure with demographic and clinical patient characteristics, CML milestones, medication toxicities, medication adherence, and germline genetic variants.

Because this is an observational study, standard-of-care therapy will not be altered during the course of participation. Blood samples will be collected at each study visit (up to 6 visits) over the course of 12 months to evaluate TKI concentrations, and PK parameters. Blood will also be collected during the first visit to isolate DNA for next generation sequencing (NGS). Demographic information will be collected at baseline, while clinical and medication adherence information will be collected at baseline and then throughout the study.

There will be no direct benefit to you for your participation. Risks are minor, but could include bruising, vein irritation, lightheadedness/dizziness, and/or infection from blood draws, as well as potential loss of confidentiality.

DETAILED DESCRIPTION:
This study is a prospective, single-institution observational study designed to evaluate associations between the pharmacokinetic (PK) parameters (e.g., clearance and exposure) for four tyrosine kinase inhibitors (TKIs) used to treat chronic phase CML with key clinical milestones in CML, as well as associations between TKI PK and medication-induced toxicities and medication adherence. The four TKIs to be evaluated in this study include bosutinib, dasatinib, imatinib, or nilotinib, while the key clinical milestones for CML include complete hematologic response (CHR) at one month, early molecular response (EMR) at 3 months and 6 months, and major molecular response (MMR) at 9 months and 12 months. A total of 150 subjects will be enrolled in the study. The enrolled study subjects will have been prescribed one of these four TKIs by a UNC medical oncologist or advanced practice provider for their diagnosed chronic phase CML. Research personnel will identify potential research subjects using data from the Carolina Data Warehouse, and pharmacy prescription claims data. Research personnel will contact patients regarding study participation in-person in clinic or over the telephone to receive informed consent.

For patients who are newly initiated on a TKI, assessment procedures will occur as close to monthly time points as possible (baseline, 1,3,6,9 12, 15, etc) with at least 30 days between draws for time points at and after 3 months. For the blood collection at 1 month, there will be a +/- 2 week window. Each patient will be enrolled in the study for a maximum of 6 different study visit days, for a total of 12 total months. If a participant changes treatment to a new TKI of interest, the participant may be followed for an additional 12 months. Active participation in the study is expected to last approximately one year for these subjects. Subjects may also be identified and enrolled after having already been initiated on TKI therapy, in which case, the duration since initiation of their TKI will be 12 total months and they will enter at the closes study time point. If enrolled subjects require a change of therapy, they will restart their participation under the new TKI at baseline and be followed for an additional 12 months. Subjects who complete the 12-month study duration and subsequently change therapy may continue participation under the new TKI and restart their participation at baseline.

All study visits will align with standard-of-care follow-up appointments such that no additional research only visits to the UNCMC are required of the subjects. Up to seventy-two hours prior to each visit, one member of the study personnel will telephone (or email, if unreachable by telephone) the subject to remind them to take their medication the days prior to their study visit, but not the day of their study visit prior to blood sample collections. Subjects will also be reminded to record the exact time and date of the two doses prior to their study visit date. Subjects may resume their normal TKI dosing regimen after completion of the study visit, at the discretion of the treating provider.

At each clinic visit, the subject will have two blood samples drawn, and will be required to complete a series of surveys (Appendices D, E). Each blood sampling will collect approximately 4mL of peripheral blood, for a total of approximately 8mL of blood per study visit. Each subject will also have an additional 4mL of blood collected once at their first study visit for DNA extraction. The first research blood sample will be collected at the beginning of the clinic visit alongside the routine blood draws and processed according to the procedures listed in Appendix C. Surveys will then be administered during the visit, and lab results and clinical data will be collected. Prior to discharge, a final research blood sample will be drawn. Phlebotomy will be performed by trained phlebotomists, nurses, or physicians in the UNCMC. Blood samples will be processed per protocol by the study personnel as trained by PI or co-investigators. A detailed summary of clinic visit procedures can be found in Appendices A and B.

For subjects enrolled on the same day as their first study visit, blood samples will be drawn at the end of the study visit. All subsequent study visits will take place as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have signed written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information
2. Patients must be ≥ 18 years old.
3. Patients must have been diagnosed with chronic phase CML.
4. Patients who will start or have already started receiving oral chemotherapy with bosutinib, dasatinib, imatinib, or nilotinib for their diagnosis of CML.

Exclusion Criteria:

1. Patients who have cognitive impairments that could affect informed decision making.
2. Patients who are prescribed bosutinib, dasatinib, imatinib, or nilotinib in combination with other chemotheapy agents (e.g., hydroxyurea or omacetaxine).
3. Patients who have undetectable BCR-ABL transcripts.
4. Patients with a confirmed T315I point mutation in BCR-ABL and/or prescribed ponatinib.
5. Patients who are incarcerated.
6. Patients with accelerated or blast phase CML.
7. Patients diagnosed with, or currently undergoing treatment for a concurrent second primary malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective, single-institution observational study is designed to evaluate associations between the pharmacokinetic (PK) parameters (e.g., clearance and exposure) for four tyrosine kinase inhibitors (TKIs) used to treat chronic phase CML with key clinical milestones in CML, as well as associations between TKI PK and medication-induced toxicities and medication adherence. The four TKIs eligible for this study include bosutinib, dasatinib, imatinib, or nilotinib. A total of 150 subjects will be enrolled in the study. The enrolled study subjects will have been prescribed one of these four TKIs by their UNC medical oncologist or advanced practice provider for their diagnosed chronic phase CML.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Correlation between TKI Exposure/Clearance and BCR-ABL transcript | 12 months
  TKI exposure/clearance will be evaluated by measuring levels of TKI in the blood during the 12 month study period. BCR-ABL transcripts at 12 months will be compared against the TKI levels.

SECONDARY OUTCOMES:
Complete Hematologic Response (CHR) | 1 month
  CHR at 1 month, defined as complete normalization of peripheral blood counts with leukocyte count < 10 x 1E9/L, platelet count < 450 x 1E9/L, no immature cells (such as myelocytes, promyelocytes, no blasts in peripheral blood, and no signs and symptoms of disease with disappearance of palpable splenomegaly.
Correlation between Early Molecular Response (EMR) and TKI Exposure/Clearance | 3 months, 6 months
  Incidence of EMR at 3 and 6 months, defined as BCR-ABL transcript ≤ 10%, will be evaluated, and will be compared against TKI levels at 3 and 6 months.
Correlation between Major Molecular response (MMR) and TKI Exposure/Clearance | 9 months, 12 months
  Incidence of MMR at 9 and 12 months, defined as BCR-ABL transcript ≤ 0.1%, will be evaluated, and will be compared against TKI levels at 9 and 12 months.
Correlation between Log10 change in BCR-ABL and TKI Exposure/Clearance | Baseline and 1, 3, 6, 9, and 12 months
  BCR-ABL transcripts will be obtained at each time point. The Log10 change in BCR-ABL transcripts will be evaluated, and will be compared against TKI levels at each time point.
Medication Adherence | Baseline and 1, 3, 6, 9, and 12 months
  Subject adherence will be evaluated at each time point during standard-of-care study visits. The Wilson's 3-item Adherence Score (WAS) tool will be administered to each subject at each visit in survey form. The WAS tool provides a score from 0-100 (0, worst; 100, best) to evaluate adherence to medications in the last 30 days.
Correlation between Medication-induced Toxicities and TKi Exposure/Clearance | Baseline and 1, 3, 6, 9, and 12 months
  Associate TKI exposure/clearance with subject-reported toxicity assessments. Medication-induced toxicity assessments will be conducted at each study visit using the validated MD Anderson Symptom Inventory for CML (MDASI-CML) tool. The MDASI-CML tool asks subjects to rate symptom severity in the last 24 hours on a 0-10 scale (0, not present; 10, as bad as one can imagine). The MDASI-CML also evaluates symptom interference with daily activities in the same manner.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Crona, PharmD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials